CLINICAL TRIAL: NCT01253577
Title: A Clinical Evaluation of a Steroid-Coated Sinus Stent When Used Following Functional Endoscopic Sinus Surgery in Patients With Chronic Sinusitis
Acronym: ADVANCE II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Intersect ENT (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P500-1009
Record Dates: First submitted 2010-12-02; First posted 2010-12-03 (Estimated); Results first posted 2015-04-13 (Estimated); Last update posted 2015-06-22 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Sinusitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Drug Coated (Active Comparator): Sinus stent coated with steroid
  Interventions: Device: Sinus Stent with drug coating
- Non coated (Placebo Comparator): Sinus stent without drug coating
  Interventions: Device: Non Coated Sinus Stent

INTERVENTIONS:
Device: Sinus Stent with drug coating — Sinus stent coated with 370 ug of the corticosteroid mometasone furoate
  Arms: Drug Coated
Device: Non Coated Sinus Stent — Sinus stent (visually identical) without drug coating
  Arms: Non coated

SUMMARY:
The purpose of this study is to assess the safety and efficacy of the Propel mometasone furoate implant when used following Functional Endoscopic Sinus Surgery (FESS) in patients with Chronic Sinusitis (CS).

DETAILED DESCRIPTION:
The purpose of this study is to assess the safety and efficacy of the Propel mometasone furoate implant when used following Functional Endoscopic Sinus Surgery (FESS) in patients with Chronic Sinusitis (CS). The Propel implant is designed to provide a mechanical spacing function within the sinus anatomy to separate mucosal tissues, provide stabilization of the middle turbinate, and thereby prevent tissue adhesions from forming. The implant is coated with a small amount of mometasone furoate (a corticosteroid) in order to help minimize post surgical inflammation within the supported tissues.

The study utilizes an intra-patient control design to assess the safety and efficacy of the drug-coated implant compared to the non-drug coated implant that is identical in appearance.

ELIGIBILITY:
Inclusion Criteria:

* Patient has bilateral chronic sinusitis confirmed by CT scan and defined as inflammation of the mucosa of the nose and paranasal sinuses of at least 8 consecutive weeks' duration.
* Patient is indicated for and has consented to FESS.
* FESS successfully completed without significant complication that in the opinion of the physician would confound study results and the patient's anatomy remains amenable to Sinus Stent placement.

CT Imaging Inclusion Criteria:

* CS diagnosis confirmed and documented by CT Scan within 6 months of the procedure.
* Patient has minimum total CT score (Lund-Mackay method) of 6. • Patient has bilateral ethmoid sinus disease confirmed by CT.

Exclusion Criteria:

* insulin dependent diabetics
* oral steroid dependent condition
* glaucoma, ocular hypertension, posterior subcapsular cataracts
* middle turbinate resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2009-12; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Marple, MD, Principal Investigator — University of Texas; Neil Bhattacharyya, MD, Principal Investigator — Brighan & Women's Hospital
Locations (11):
- United States (11):
  - Central California ENT, Fresno, California
  - Colorado ENT & Allergy, Colorado Springs, Colorado
  - Northwestern University, Chicago, Illinois
  - Northshore University Health System, Evanston, Illinois
  - Advanced ENT & Allergy, Louisville, Kentucky
  - Charlotte Eye, ENT Associates, Charlotte, North Carolina
  - Austin ENT Clinics, Austin, Texas
  - University of Texas SW Medical School, Dallas, Texas
  - University of Texas Medical School, Houston, Texas
  - Intermountain ENT, Salt Lake City, Utah
  - Eastern Virgina Medical School, Norfolk, Virginia

REFERENCES:
- [Result] Han JK, Marple BF, Smith TL, Murr AH, Lanier BJ, Stambaugh JW, Mugglin AS. Effect of steroid-releasing sinus implants on postoperative medical and surgical interventions: an efficacy meta-analysis. Int Forum Allergy Rhinol. 2012 Jul-Aug;2(4):271-9. doi: 10.1002/alr.21044. Epub 2012 May 1. PMID 22550039

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited in the United States between December 2009 and July 2010 from eleven otolaryngology-head and neck surgery centers by 31 surgeons representing both academic and private practices.
Pre-assignment Details: Sinus randomization was performed at the end of successful endoscopic sinus surgery.
Groups:
- Sinus Stent: Participants sinuses were randomized to receive drug-coated sinus stent on one side and non-drug coated control stent on the contralateral side in a split-face design.
Period: Overall Study
Arm/Group | Sinus Stent
Started | 105
Completed | 102
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Sinus Stent
Number analyzed (Participants) | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 95
  >=65 years | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 60
Region of Enrollment [Number; unit: participants]
  United States | 105

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Sinuses Requiring Post-operative Intervention
Description: Post-operative interventions include either need for surgical adhesion lysis or the need for oral steroids prescription, as determined from video-endoscopies reviewed by a panel of independent blinded sinus surgeons.
Time Frame: 30-days
Population: All 105 subjects were present for the primary endpoint exam. However n=96 is the number of subjects where both sinus sides had video-endoscopies able to be graded by the independent panel.
Measure: Mean (95% Confidence Interval); unit: percentage of sinuses
Groups:
- Drug-Coated Implant Side: Sinus stent coated with steroid
- Non-coated Implant Side: Sinus stent without drug coating
Arm/Group | Drug-Coated Implant Side | Non-coated Implant Side
Number analyzed (Participants) | 96 | 96
percentage of sinuses | 33.3 [24.0 to 43.7] | 46.9 [36.6 to 57.3]
Statistical Analysis 1: Comparison: Drug-Coated Implant Side vs Non-coated Implant Side; Test type: Superiority or Other; p = 0.0280, McNemar

2. Primary Outcome: Percentage of Patients With Clinically Significant Increase in Intra-ocular Pressure
Description: clinically significant IOP elevation is a change from baseline of >10 mm Hg on sinus side with drug-coated implant but not on side with control implant
Time Frame: 90 days
Population: Two patients did not have their ocular exam performed at day 90 (LTFU) but had ocular exams at earlier time points.
Measure: Mean (95% Confidence Interval); unit: percentage of patients
Arm/Group | All Subjects
Number analyzed (Participants) | 103
percentage of patients | 0 [0 to 3.52]
Statistical Analysis 1: Comparison: All Subjects; Test type: Superiority or Other; p < 0.0001, Fisher Exact

3. Secondary Outcome: Percentage of Sinuses That Developed Frank Polyposis
Description: Frank polyposis means polyps grade 2 or 3, which was determined from video-endoscopies reviewed by a panel of independent blinded sinus surgeons.
Time Frame: 30 days
Population: All 105 subjects were present for this endpoint exam. However n=85 is the number of subjects where both sinus sides had video-endoscopies able to be graded by the independent panel.
Measure: Mean (95% Confidence Interval); unit: percentage of sinuses
Arm/Group | Drug-Coated Implant Side | Non-coated Implant Side
Number analyzed (Participants) | 85 | 85
percentage of sinuses | 18.8 [11.2 to 28.8] | 34.1 [24.2 to 45.2]
Statistical Analysis 1: Comparison: Drug-Coated Implant Side vs Non-coated Implant Side; Test type: Superiority or Other; p = 0.0023, McNemar

ADVERSE EVENTS:
Time Frame: 3 Months
Groups:
- All Patients: Patients served as their own controls in the study, with a drug-coated stent placed on one sinus side and a non-drug-coated control placed on contralateral side. Therefore adverse events are listed for the entire 105-patient cohort rather than by treatment group.
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 0/105
Other Adverse Events (participants affected / at risk) | 45/105
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=105)
Headache (Nervous system disorders) | 5 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Bronchitis (Infections and infestations) | 3 (3)
Sinusitis (Infections and infestations) | 34 (34)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less